CLINICAL TRIAL: NCT00312390
Title: Amblyopia and Neurovascular Coupling in the Retina of Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhöfer, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-070503
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Amblyopia; Regional Blood Flow
Keywords: Amblyopia; Retinal vessel diameters; Retinal blood flow; Flicker
MeSH Terms: conditions — Amblyopia; photopsia | interventions — Flicker Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Control Subjects (Other)
  Interventions: Procedure: Flicker; Procedure: Retinal Vessel Diameter; Procedure: Retinal Blood Flow
- Subjects with amblyopia (Other)
  Interventions: Procedure: Flicker; Procedure: Retinal Vessel Diameter; Procedure: Retinal Blood Flow

INTERVENTIONS:
Procedure: Flicker
Procedure: Retinal Vessel Diameter
Procedure: Retinal Blood Flow

SUMMARY:
The visual disorder of amblyopia affects 2% to 3% of the population. Amblyopia is a developmental condition that is characterized by reduced vision of the eye due to the presence of a sensory impediment during visual development, such as strabismus (ocular misalignment) or anisometropia (unequal refractive error), occurring early in life. Recent studies in humans and animals point towards a cortical locus for the processing deficit in amblyopia, revealing sensory deficits at the signal cell level that include reduced spatial resolution, reduced contrast sensitivity, and a reduced number of binocular neural cells. In the retina, however, no abnormalities have yet been reported.

Like in the brain blood flow in the retina is coupled to neuronal activity. This phenomenon has been measured by different study groups with non invasive techniques in the brain and retina. We therefore use a Zeiss fundus camera for the assessment of retinal vessel diameters. This so called retinal vessel analyzer (RVA) is a combination of a fundus camera connected to a high resolution video camera equipped with a software based analyzing system. An unprecedented reproducibility and sensitivity of retinal vessel diameter measurements is attained with this system. In addition this system allows real time analysis of retinal vessels as well as off-line determinations from video tape. A special provocation test, which minimizes risk and discomfort to the subject under study is applied through the illumination pathway of the fundus camera: Diffuse luminance flicker is used as a stimulus to augment intrinsic mechanisms by which the retina can vary the vascular supply, in correspondence with local variations of functional activity. This system allows to study the flicker response of retinal vessels, which is within a magnitude of 6 to 8%.

However, the exact mechanisms underlying this phenomenon are not fully understood. Especially in the eye it is not clear whether it is an exclusive metabolic effect within the retina and the surrounding blood vessels or dependent of central regulatory brain functions.

The purpose of the current study is to improve our understanding of the mechanisms underlying flicker evoked responses of retinal blood vessels in humans. It is not clear whether the retina of amblyopic eyes can regulate retinal blood flow in response to increased metabolic demands as induced during flicking light stimulation. A detail understanding of the metabolic and functional processes within the retina of patients with amblyopia is a prerequisite for further research to prevent amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for healthy subjects:
* Women and men, aged between 18 and 60 years
* Matched with regard to age, sex and smoking status
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia of less than 3.0 dpt
* Inclusion criteria for patients with amblyopia as a result of anisometropia or strabismus:
* Normal ophthalmic findings except amblyopia on one eye resulting from anisometropia or strabismus with a visual acuity between log Mar 0.3 and 0.7 (Snellen 0.2-0.5) with best correction on the amblyopic eye and 0.1 (Snellen 0.9) or better on the contralateral eye
* Anisometropia of more 3 dpt (patients with anisometropia)
* Women and men, aged between 18 and 60 years
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* pregnancy
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2003-07

PRIMARY OUTCOMES:
Retinal vessel diameter | 10 minutes
Time course of diameter changes induced by flicker light stimulation | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria